CLINICAL TRIAL: NCT01900834
Title: An Observational Study Evaluating Biomarker Expression in Diabetic and Healthy Subjects Over a One Year Period
Brief Title: Evaluation of Biomarker Expression in Diabetic and Healthy Subjects Over a One Year Period
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4099; U1111-1140-1650 (Other: WHO)
Record Dates: First submitted 2013-06-28; First posted 2013-07-17 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Monthly venous blood samples within the first half year and thereafter bi-monthly the rest of the year. A subgroup of the subjects will also be invited for a visit within a week after the former visit to assess the variation of the biomarkers within a week. The blood samples will be assayed for peripheral blood mononuclear cells (PBMC) specificity, phenotype and function as well as for islet autoantibodies (presence and precise titers), for autoantibody isotypes and diabetes risk parameters. Finally C-peptide levels and residual beta cell function will be measured three times during the study after a mix meal tolerance test (MMTT) in subjects with T1D.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — The participants will not receive any treatment

SUMMARY:
This study is conducted in the United States of America (USA). The aim of this study is to assess longitudinal variation of immune biomarkers in subjects with type 1 diabetes (T1D), type 2 diabetes (T2D) and healthy, non-diabetic subjects over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* T1D
* Male or female subjects diagnosed within the last 3 years and with good general health based on medical history
* Age above or equal to 14 years and below or equal to 40 years
* Body weight above 45 kg
* T2D
* Male or female subjects diagnosed within the last 15 years with good general health based on medical history
* HbA1c between 6.5% and 10%
* Body mass index (BMI) below 45 kg/m^2
* Age above or equal to 18 and below 65 years
* On insulin treatment
* HS
* Male or female subjects with good general heath based on medical history
* Age above or equal to 18 years and below or equal to 40 years

Exclusion Criteria:

* Any chronic disorder (besides T1D or T2D) or severe disease which, in the opinion of the investigator, might jeopardize subject's safety or compliance with the protocol
* Female of child-bearing potential who is pregnant, breast-feeding, or intends to become pregnant

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects with T1D, T2D and healthy subjects (HS) without personal or first degree family history of autoimmunity of diabetes. The HS will be mean age-matched with the T1D subjects.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Variation in CD8 (cluster of differentiation) +T-cell specificity profiling | Over a one year period

SECONDARY OUTCOMES:
Variation in CD4 +T-cell specificity profiling | Over a one year period
Change in stimulated C-peptide | Baseline, one year
Fluctuation in islet autoantibodies titers | Over a one year period
Variation in HbA1c (glycosylated haemoglobin) | Over a one year period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com